CLINICAL TRIAL: NCT04608929
Title: The Effect of Kegel Exercise-focused Interventions on Urinary Incontinence in Elderly Women
Brief Title: Kegel Exercise-focused Interventions in Elderly Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Hilal Gamze Hakbilen, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Akdeniz Uni
Record Dates: First submitted 2020-10-21; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Urinary Incontinence; Kegel Exercises; Nursing
MeSH Terms: conditions — Urinary Incontinence | interventions — House Calls

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The arm where the Kegel exercise focused intervention is applied
  Interventions: Behavioral: Kegel exercise-focused interventions
- Control (Experimental): The arm where home follow-up and scale evaluations are made
  Interventions: Other: Home visit and scale evaluations

INTERVENTIONS:
Behavioral: Kegel exercise-focused interventions — After the patients in the intervention group were interviewed on the telephone, the second home visit. During this visit, the patients were trained on Kegel exercises and they were administered the ICIQ-SF. Six weeks after the second visit, the third home visit was paid to determine whether the patients did the Kegel exercises and whether they did them accurately, to assess the perceived impact and to re-administer the ICIQ-SF. After the 2nd and 3rd visit, the patients were called once a week for 6 weeks to monitor if they kept up with doing the Kegel exercises as they were taught. Six weeks later, the 4th home visit were paid to the patients. During this visit, whether the patients did the Kegel exercises and whether they did them accurately was determined, the perceived impact was assessed and the ICIQ-SF was re-administered.
  Arms: Intervention
Other: Home visit and scale evaluations — After the 1st visit, the patients included in the control group were called by phone and the 2nd home visit was planned. During the second home visit, the ICIQ-SF was administered to them. At the 3rd home visit paid 6 weeks after the 2nd visit, the ICIQ-SF was re-administered to the patients and the perceived impact assessment was performed. During the 4th home visit paid 6 weeks after the 3rd home visit, the ICIQ-SF was re-administered to the patients, assessment of the perceived impact was performed, and finally they were given training on Kegel exercises.
  Arms: Control

SUMMARY:
Purpose: This study was conducted to investigate the effects of Kegel exercises-focused intervention undergone by elderly women diagnosed with urinary incontinence on their incontinence, quality of life and perceived impact level.

Design: The study has a single-blind randomized controlled experimental research design.

Methods: The study was carried out between December 2017 and March 2019 with 60 elderly women registered at the Home Health Unit of a Metropolitan Municipality in Turkey. The women were assigned to the intervention (n=30) and control (n=30) groups. The participants in the intervention group were paid home visits to provide them with individual training and counseling on Kegel exercises. Whether the participants did the exercises was followed up by weekly phone calls. The frequency of urinary incontinence, the amount of urine leaking and the quality of life of the participants and their complaints about incontinence were assessed with the International Consultation on Incontinence Questionnaire Short Form and questions on the assessment of the perceived impact at the onset of the study (0th week), and at home visits paid at the 6th and 12th weeks after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 65,
* Being women,
* Diagnosed with UI,
* Being literate,
* Being able to communicate in Turkish,
* Standardized Mini Mental Test result was > 24,
* Agree to participate in research.

Exclusion Criteria:

* Who had received training on incontinence and Kegel exercises in the last 1 year,
* Had symptoms of urinary tract infection were identified,
* Being treated for UI,
* Having health problems affecting the muscle and nervous system,
* Being not able to perform daily life activities,
* Having pelvic organ prolapse,

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Change in frequency of urinary incontinence after onset | 6. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Change in frequency of urinary incontinence after onset | 12. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Change in amount of urinary incontinence after onset | 6. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Change in amount of urinary incontinence after onset | 12. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Change in effects of urinary incontinence on daily life after onset | 6. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Change in effects of urinary incontinence on daily life after onset | 12. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Change in assessment of the perceived impact after onset | 6. week
  Patient Information Form developed by the researchers based on the pertinent literature consists of 5 parts and 28 questions. The first part questions the patient's age, height, weight etc. The second part is on the patient's obstetric characteristics. The third part questions the patient's health history. The fourth part questions the patient's incontinence status. The fifth part is on the assessment of the perceived impact.
Change in assessment of the perceived impact after onset | 12. week
  Patient Information Form developed by the researchers based on the pertinent literature consists of 5 parts and 28 questions. The first part questions the patient's age, height, weight etc. The second part is on the patient's obstetric characteristics. The third part questions the patient's health history. The fourth part questions the patient's incontinence status. The fifth part is on the assessment of the perceived impact.

SECONDARY OUTCOMES:
Evaluation of the participants in terms of performing Kegel Exercises | 6. week
  The Weekly Exercise Follow-up Form was developed by the researchers to assess the frequency of exercises in patients who were given Kegel exercise training. The Weekly Exercise Follow-up Form has a timetable consisting of 7 days of the week and 3 parts of the day (morning, noon and evening). The patients mark the timetable by placing an "X" on the blank corresponding to the time when they perform the exercise.
Evaluation of the participants in terms of performing Kegel Exercises | 12. week
  The Weekly Exercise Follow-up Form was developed by the researchers to assess the frequency of exercises in patients who were given Kegel exercise training. The Weekly Exercise Follow-up Form has a timetable consisting of 7 days of the week and 3 parts of the day (morning, noon and evening). The patients mark the timetable by placing an "X" on the blank corresponding to the time when they perform the exercise.
Assesment of which cases do you leak urine? | 6. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.
Assesment of which cases do you leak urine? | 12. week
  The International Consultation on Incontinence Questionnaire Short Form has the following four sub-dimensions: frequency of urinary incontinence, the amount of leakage, the impact of urinary incontinence on daily life, and causes of urinary incontinence. The first three sub-dimensions are included in scoring. The responses given to the fourth dimension, which is not included in the scoring process enable the health professional to determine the type of urinary incontinence based on the person's complaints. The minimum and maximum possible scores to be obtained from the scale are 0 and 21 respectively. While low scores indicate that urinary incontinence has little impact on the quality of life, high scores indicate that urinary incontinence has a great impact on the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Home Health Unit of Antalya Metropolitan Municipality, Antalya, Muratpaşa, Turkey (Türkiye)